CLINICAL TRIAL: NCT04821739
Title: A Prospective Multi-Center Study of the AGN1 Local Osteo-Enhancement Procedure (LOEP) SV Kit in Patients With Vertebral Compression Fractures (VCFs)
Brief Title: RISE - Study of the AGN1 LOEP SV Kit in Patients With Vertebral Compression Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AgNovos Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGN-CIP-200
Record Dates: First submitted 2021-03-11; First posted 2021-03-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Vertebral Compression Fracture; Vertebral Compression; Vertebral Fracture
Keywords: LOEP; AGN1; RISE; Local Osteo-Enhancement Procedure
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with AGN1 LOEP SV Kit (Experimental): VCF is treated with the AGN1 LOEP SV Kit
  Interventions: Device: AGN1 LOEP SV Kit

INTERVENTIONS:
Device: AGN1 LOEP SV Kit — The AGN1 LOEP SV Kit is intended for fixation of pathological fractures of the vertebral body using vertebral augmentation.

SUMMARY:
This study is a prospective, single-arm, multi-center, European clinical study designed to evaluate the clinical performance and safety of the AGN1 LOEP SV Kit for the treatment of painful VCFs.

DETAILED DESCRIPTION:
A maximum of 100 subjects will be treated at up to 10 study sites across Europe. Follow up visits will be conducted at 1 day, 1 month, 3 months, 12 months and 24 months after the procedure.

Study enrollment will occur in three stages:

Stage 1: 5 subjects to evaluate safety at 3 months Stage 2: 30 subjects to evaluate safety at 3 months Stage 3: 100 subjects to evaluate safety and performance at 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female 50 years of age or older at time of study treatment.
2. Criterion omitted
3. Subject has only one (1) acute VCF. Subjects are eligible if they have an asymptomatic healed VCF at any non-target vertebral level.
4. This VCF meets all of the following criteria:

   1. Fracture due to diagnosed or presumed underlying osteoporosis
   2. VCF from T1 to L5 inclusive
   3. Fracture age ≤6 months at time of treatment
5. Target VCF shows loss of height in the anterior or middle portion of the vertebral body of not more than 50% based on X-ray at baseline.
6. Target VCF is acute or persistent (not healed), as demonstrated by T2 weighted STIR MRI, bone scan, CT, serial radiographs, or other imaging demonstrating acuity.
7. Subject has central pain upon palpation over the spinal process at the target vertebral body.
8. Subject has failed conservative medical therapy, defined as either having a VAS back pain score of ≥ 70 mm after 24 hours to 6 weeks of conservative care or a VAS back pain score of ≥ 50 mm after 6 weeks of conservative care.
9. Subject has an Oswestry Disability Index (ODI) score of ≥ 30%.
10. Subject is capable of giving written informed consent to participate in the study.
11. The subject's willingness, ability, and commitment to participate in screening, treatment, and all follow-up evaluations for the full length of the study has been documented.

Exclusion Criteria:

1. Target VCF is due to underlying or suspected tumor.
2. Target VCF is due to high-energy trauma.
3. Target VCF is diagnosed as an osteonecrotic fracture.
4. Target VCF has segmental kyphosis of > 30°.
5. Target VCF is unstable including split or burst fractures.
6. Subject has had any prior surgical treatment at the target VCF or adjacent vertebral level (above or below VCF).
7. Subject has neurologic symptoms, deficits, or radiculopathy related to the VCF.
8. Subject has spinal canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression at the level to be treated.
9. Subject has pain based on clinical diagnosis of herniated nucleus pulposus or severe spinal stenosis (progressive weakness or paralysis).
10. Subject has spondylolisthesis > Grade 1 at target vertebral body.
11. Subject has pain due to any other condition that requires daily narcotic medication.
12. Subject has severe cardiopulmonary deficiencies.
13. Subject has a bleeding disorder.
14. Subject has a Body Mass Index (BMI) > 35.
15. Subject has a history of metabolic bone disease other than osteoporosis (e.g., Paget's disease, renal osteodystrophy, or osteomalacia).
16. Subject has a history of tuberculosis spondylitis.
17. Subject has a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for five (5) years.
18. Subject is on oral or parenteral immune-suppressive drugs.
19. Subject has an active bone infection at target VCF.
20. Subject has uncontrolled diabetes mellitus, as determined by the judgment of the Investigator.
21. Subject has severe renal insufficiency defined as an estimated glomerular filtration rate (eGFR) < 30 mL/min.
22. Subject has a diagnosed calcium metabolism disorder.
23. Subject has known allergies to calcium-based bone void fillers.
24. Subject is pregnant or planning to become pregnant during participation in the study.
25. In the judgment of the Investigator, the subject is not a good study candidate (e.g., inability to maintain follow-up schedule, comorbidity or poor general physical/mental health, or drug or alcohol abuse issues).
26. Subject is currently enrolled in another interventional clinical study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Back Pain from Baseline | 12 months
  Change in Back Pain at 12 months from Baseline as indicated by Visual Analogue Scale (VAS), measured on a continuous 100 mm line.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Arab Motlagh, MD, Principal Investigator — Sana Klinikum Offenbach GmbH
Locations (4):
- Germany (2):
  - Orthopedic University Hospital Friedrichsheim, Frankfurt am Main, Hesse
  - Sana Klinikum Offenbach GmbH, Offenbach
- Spain (2):
  - Hospital Clinico Universitario de Valladolid, Valladolid, Valladolid
  - Vall d'Hebron University Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: No